CLINICAL TRIAL: NCT06240637
Title: Telemonitoring Utility in the Process of Adaptation to Home Mechanical Ventilation
Brief Title: Telemonitoring Utility in the Process of Adaptation to Home Mechanical Ventilation (HMV)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Societat Catalana de Pneumologia (SOCAP) (Unknown); Sociedad Española de Neumología y Cirugía Torácica (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIBSP-TEL-2022-132
Record Dates: First submitted 2024-01-17; First posted 2024-02-05 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-01

CONDITIONS: Non Invasive Ventilation
Keywords: Telemonitoring; NIV

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemonitoring group (Active Comparator): Follow-up model adding telemonitoring with remote review of HMV data on a daily basis during the first 2 weeks and subsequently weekly up to 6 months. Telephone contact with the patient in case of any eventuality and timely adjustments to therapy. Patients will attend in-person follow-up visits at 2, 4, and 6 months after initiating HMV. Clinical and gasometric control, nocturnal pulse oximetry, questionnaires, and download of ventilator data. Timely adjustments to therapy.
  Interventions: Other: Telemonitoring
- Control group (No Intervention): Exclusive in-person follow-up model with control visits at 2 weeks, 1, 2, 4, and 6 months after initiating HMV. Clinical and gasometric control, nocturnal pulse oximetry, questionnaires, and download of ventilator data. Timely adjustments to therapy

INTERVENTIONS:
Other: Telemonitoring — A networked platform that enables the telemonitoring of both compliance data and the patient's ventilatory pattern, allowing the assessment of flow/pressure curves as well as leaks or events related to the upper airway.
  Arms: Telemonitoring group

SUMMARY:
The goal of this clinical trial is to evaluate whether telemonitoring, added to the usual process of adaptation to home mechanical ventilation (HMV), achieves a more efficient correction of hypoventilation (reduction of hypercapnia).

DETAILED DESCRIPTION:
The study population consist of patients with hypercapnic respiratory failure eligible for Home Mechanical Ventilation (HMV) with a total of 48 subjects (24 per group).

In those patients with hypercapnic respiratory failure who have an indication for home mechanical ventilation (HMV), without criteria for life support, the initial titration will be performed following the protocol of the Pulmonology Service. After their education, patients will be randomized into one of the following groups: the control group and the telemonitoring group with daily review of Home Mechanical Ventilation (HMV) data. The objectives are to evaluate whether hypoventilation is corrected more efficiently, compare treatment adherence between both groups, analyze unforeseen visits, and assess the number of hospital admissions.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hypercapnic respiratory failure with indication for home mechanical ventilation.
* Patients who require ventilation with spontaneous-timed mode.
* Signing of informed consent.

Exclusion Criteria:

* Patient already treated with mechanical ventilation or home CPAP.
* Patient requiring mechanical ventilation as life support.
* Pregnancy.
* Cognitive impairment that makes it impossible to understand the informed consent for the study.
* Psychiatric pathology that makes compliance with therapy or its follow-up difficult.
* Impossibility of complying with the protocol.
* Expected survival less than 12 months.
* Any other condition that, in the opinion of the researcher, could interfere with the objectives of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-02-17 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of pCO2 by arterial blood gas | 6 months
  The partial pressure of carbon dioxide (PCO2) is the measure of carbon dioxide within arterial or venous blood. The moment (day) in which normal pCO2 is detected (pCO2 < 45 mmHg) will be determined as the success of the therapy.

SECONDARY OUTCOMES:
Adherence | 6 months
  Compare treatment adherence with Home Mechanical Ventilation (HMV) between monitoring with and without telemonitoring.
Unforeseen visits | 6 months
  Compare the number of unforeseen visits generated with both systems.
Hospital admissions | 6 months
  Compare the number of hospital admissions due to acute exacerbation of chronic respiratory failure with both adaptation systems.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

DOCUMENTS (1):
  • Informed Consent Form (2023-07-28): https://cdn.clinicaltrials.gov/large-docs/37/NCT06240637/ICF_000.pdf